CLINICAL TRIAL: NCT01293747
Title: Multiple-dose Pharmacokinetic Study of Two Aqueous Suspensions of Estradiol and Progesterone Microspheres (1 mg/20 mg & 0.5 mg/15 mg) for Intramuscular Administration, in Postmenopausal Volunteers.
Brief Title: Pharmacokinetics of Injectable Estradiol and Progesterone Microspheres Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Productos Científicos S. A. de C. V. (Industry)
Responsible Party: Principal Investigator, Roberto Bernardo Escudero, Principal Investigator, Productos Científicos S. A. de C. V.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0903/I/PRO
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Menopause
Keywords: Estrogen; Progesterone; Microspheres; Menopause; Pharmacokinetics
MeSH Terms: interventions — Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estradiol 0.5 mg/Progesterone 15 mg microspheres (Experimental): Estradiol 0.5 mg and progesterone 15 mg microspheres injectable aqueous suspension
  Interventions: Drug: Estradiol + Progesterone
- Estradiol 1 mg/Progesterone 20 mg microspheres (Experimental): Estradiol 1 mg and progesterone 20 mg microspheres injectable aqueous suspension
  Interventions: Drug: Estradiol + Progesterone

INTERVENTIONS:
Drug: Estradiol + Progesterone — Estradiol 1 mg and progesterone 20 mg microspheres injectable aqueous suspension, intramuscular monthly injection for a total of 4 doses.
  Arms: Estradiol 1 mg/Progesterone 20 mg microspheres
Drug: Estradiol + Progesterone — Estradiol 0.5 mg and progesterone 15 mg microspheres injectable aqueous suspension, intramuscular monthly injection for a total of 4 doses.
  Arms: Estradiol 0.5 mg/Progesterone 15 mg microspheres

SUMMARY:
Phase I pharmacokinetic study

Main objective:

To determine plasmatic profiles and pharmacokinetic parameters of estradiol and progesterone on each of the formulations studied, after multiple-dose administration

Study design:

Randomized, controlled, open-label, parallel, pharmacokinetic study

Sites: 1

Subjects: 30 postmenopausal women

DETAILED DESCRIPTION:
Sites: 1

Phase: 1

Main objective:

To determine plasmatic profiles and pharmacokinetic parameters of estradiol and progesterone on each of the formulations studied, after multiple-dose administration.

Secondary objectives:

To determine bioavailability of each of the formulations studied, after multiple-dose-administration. Describe tolerability of each of the formulations studied, after multiple-dose administration.

Study design: Randomized, controlled, open-label, parallel, pharmacokinetic study

Investigational Products:

* Estradiol and progesterone microspheres aqueous suspension (1 mg/20 mg)
* Estradiol and progesterone microspheres aqueous suspension (0.5 mg/15 mg)

Study subjects: 30 postmenopausal women 45 - 65 years old

Brief description: After written informed consent, 30 eligible women will be randomized to study treatments (one IM injection each 28 days, for a total of 4 doses). Blood samples will be obtained for pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 45 to 65 years old
* Able to read and write
* Postmenopausal
* Body Mass Index equal or below 34.99 kg/m2
* Healthy
* Normal uterus
* Time availability

Exclusion Criteria:

* Hypersensitivity to progesterone or related compounds
* Hypersensitivity to estrogens
* Hysterectomy
* History or present hormone-dependent tumor
* History or present uterine cervix dysplasia
* Abnormal and clinically-significant laboratory test results
* Family history of breast cancer
* History of thromboembolic disease
* Non-controlled hypertension
* History of stroke
* History of cardiac valve surgery
* Renal failure
* Hepatic failure
* Non-controlled diabetes
* History of serious neurologic disease
* Reduced mobility
* Anemia
* Previous or concomitant hormone therapy
* Previous or concomitant therapy with inhibitors or inductors of cytochrome

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 0 - 60 Days
  Estrogen and progesterone plasma concentrations and pharmacokinetic parameters.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 0 - 60 days
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability. Adverse events will be evaluated through periodic clinical evaluations and laboratory tests (comparison between enrollment and discharge).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bernardo, MSc, Principal Investigator — Asociación Mexicana para la Investigación Clínica, A. C. (AMIC)
Locations (1):
- Asociación Mexicana para la Investigación Clínica, A. C. (AMIC), Pachuca, Hidalgo, Mexico